CLINICAL TRIAL: NCT04919694
Title: The Therapeutic Effect of Combination of Orbital Compression Surgery and Strabismus Surgery in Patients With Moderate to Severe Thyroid Associated Ophthalmopathy
Brief Title: Combination of Orbital Compression Surgery and Strabismus Surgery for Thyroid Associated Ophthalmopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huasheng Yang, Sun Yat-sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: yanghs20210106
Record Dates: First submitted 2021-01-19; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Thyroid Associated Ophthalmopathy
MeSH Terms: conditions — Graves Ophthalmopathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combination of orbital compression and strabismus surgery (Experimental): orbital compression and strabismus surgery are performed at the same time
  Interventions: Procedure: combination of orbital compression surgery and strabismus surgery
- perform strabismus surgery after orbital compression (Active Comparator): Firstly, perform orbital compression, after about 3 to 6 months ,strabismus surgery is done.
  Interventions: Procedure: orbital compression

INTERVENTIONS:
Procedure: combination of orbital compression surgery and strabismus surgery — combination of orbital compression surgery and strabismus surgery at the same time
  Arms: combination of orbital compression and strabismus surgery
Procedure: orbital compression — orbital compression
  Arms: perform strabismus surgery after orbital compression

SUMMARY:
The purpose of this study is to determine whether combination of orbital compression surgery with strabismus surgery is better than strabismus surgery after orbital compression surgery in the treatment of moderate-to-severe thyroid associated ophthalmopathy

DETAILED DESCRIPTION:
This study will be a interventional case series. Patients with moderate-to-severe thyroid associated ophthalmopathy will be randomized to receive combination of orbital compression surgery with strabismus surgery or strabismus surgery after orbial compression surgery.Patients will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* moderate-to-severe thyroid associate ophthalmopathy
* CAS≤3 score
* monocular strabismus,deviation≥20° or 35▲
* stable thyroid function for at least 6 months, confirmed by an endocrinologist

Exclusion Criteria:

* any previous disease in the study eye.
* any previous systematic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
quality of life ,measured by GO-QoL(quality of life with Grave's Orbitopathy) . | 6 weeks after surgery
  All GO-QoL questions were scored as 'severely limited' (one point), 'a little limited' (two points) or 'not limited at all' (three points). The questions 1-8 for visual functioning (VF) and questions 9-16 for appearance (AP)were summed to produce two raw scores from 8 to 24 points and then transformed to two total scores from 0 to 100 by the following formula: total score = [(raw score - 8)/16 9 100]. In both cases, higher total scores indicate better QoL. When there were missing values, total scores were calculated for the remaining completed items. The transformation was then adjusted to total score = [(raw score - *)/(2x*) x100] where * is the number of completed items.
quality of life, measured by GO-QoL(quality of life with Grave's Orbitopathy) . | 6 months
  All GO-QoL questions were scored as 'severely limited' (one point), 'a little limited' (two points) or 'not limited at all' (three points). The questions 1-8 for visual functioning (VF) and questions 9-16 for appearance (AP)were summed to produce two raw scores from 8 to 24 points and then transformed to two total scores from 0 to 100 by the following formula: total score = [(raw score - 8)/16 9 100]. In both cases, higher total scores indicate better QoL. When there were missing values, total scores were calculated for the remaining completed items. The transformation was then adjusted to total score = [(raw score - *)/(2x*) x100] where * is the number of completed items.

SECONDARY OUTCOMES:
strabismus status | 6 weeks after surgery
  angle of deviation including up-gaze, down-gaze ,left and right-gaze
strabismus status | 6 months after surgery
  angle of deviation including up-gaze, down-gaze ,left and right-gaze

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China